CLINICAL TRIAL: NCT05957185
Title: Effects of Oral Microbial Protease Supplementation on Postprandial Plasma Amino Acid Concentrations and Appetite in Healthy Adults: A Randomized, Double-Blind, Placebo-Controlled, Crossover Clinical Trial
Brief Title: Effects of Microbial Protease Supplementation on Postprandial Plasma Amino Acid Concentrations and Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BIO-CAT, Inc. (Industry)
Collaborators: McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BCCT-TACV-0010; A05-M24-23A (Other: McGill University)
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Digestive Health; Gastrointestinal Health; Appetitive Behavior
Keywords: protease; digestive enzyme; digestion; dietary supplement
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P3 - WHEY (Active Comparator): OPTIZIOME® P3 HYDROLYZER® - WHEY (P3 - WHEY) is a mixture of 3 microbial protease preparations with 50,000 HUT fungal proteolytic activity units per 250 mg dose.
  Interventions: Dietary Supplement: OPTIZIOME® P³ HYDROLYZER® - WHEY
- Placebo (Placebo Comparator): Maltodextrin from waxy maize at 265 mg per dose.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: OPTIZIOME® P³ HYDROLYZER® - WHEY — One dose of P3 - WHEY will be combined with 31.9 grams whey protein concentrate in 300 mL water and consumed within 5 minutes at the start of each of the aminoacidemia trials.
  Other Names: P3 - WHEY; P3 HYDROLYZER® - WHEY
  Arms: P3 - WHEY
Other: Placebo — One dose of placebo maltodextrain will be combined with 31.9 grams whey protein concentrate in 300 mL water and consumed within 5 minutes at the start of each of the aminoacidemia trials.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to assess the effect of co-ingestion of microbial proteases and whey protein concentrate (WPC) on postprandial plasma amino acid concentrations in healthy adult participants compared to WPC with placebo. The secondary purpose is to assess the effect of co-ingestion of microbial proteases and WPC on postprandial glycemic response, subjective appetite sensations, gut-derived appetite regulating hormones, ad libitum meal intake, and gastrointestinal tolerability in healthy adult participants compared to WPC with placebo.

DETAILED DESCRIPTION:
A within-subject crossover design will be used for this randomized, double-blind, placebo-controlled study in health adults to assess the efficacy of a microbial protease mixture (from Aspergillus species) on enhancing postprandial aminoacidemia after consumption of a whey protein shake. There are two treatment groups in this crossover trial, including one microbial protease group and one placebo group. A total of 24 participants will be enrolled and undergo both treatment phases with a minimum 7-day washout.

The study will last no less than 8 days and up to 72 days for each participant, including screening, washout, and end of study (EOS) visit. The study will include a screening visit (Visit 1) followed by a screening period lasting up to 30 days, the phase 1 aminoacidemia trial on Day 1 (Visit 2), minimum 7-day washout with a window of +35 days, followed by the phase 2 aminoacidemia trial (EOS Visit 3, Day 8 +35 days).

During the aminoacidemia trials, participants will arrive to the clinic in a fasted state, and 31.9 grams whey protein concentrate (WPC) in 300 mL water with microbial proteases or placebo will be administered. Blood will be collected at baseline and 11 postprandial timepoints across 4 hours for plasma amino acid, glucose, and insulin quantitation. Blood will also be utilized for quantitation of the anorexigenic, satiety-related peptide hormones glucagon-like peptide 1 (GLP-1) and peptide YY (PYY), and the orexigenic peptide hormone ghrelin.

Additionally, changes in appetite sensations will be assessed by visual analog score (VAS) responses to 5 questions at baseline, directly after consumption of study products, and postprandially every half hour. Palatability of the study products will be assessed by 5-item Palatability Questionnaire. Gastrointestinal tolerability will be assessed by 8-item modified Gastrointestinal Tolerance Questionnaire (mGITQ) at the end of the 4-hour aminoacidemia trial.

To further investigate appetite and satiety, an test meal will be provided at 4 hours for the determination of energy intake, followed by a final appetite VAS questionnaire immediately after the test meal. The maximum time to finish the test meal is 30 minutes.

To account for the potential influence of menstrual cycle timing on the outcomes of interest, female subjects will be instructed to contact the clinic on day 1 of their menses so that Visit 2 (Day 1) can be scheduled at the end of menses, but still during the follicular phase of their menstrual cycle. The follicular phase is defined as days 1-14, where day 1 is the first day of menses. Therefore, Visit 2 (Day 1) and Visit 3 for female participants will occur approximately 3-5 days after start of menses, but on or before day 14 of the follicular phase (+4 day window), unless Visit 3 can be scheduled within the same follicular phase as Visit 2, with an at least 7-day washout.

The study will include a total of three in-person visit days: screening (Visit 1), phase 1 (Visit 2), and phase 2/EOS (Visit 3). Study endpoints include postprandial plasma amino acid concentrations, postprandial plasma glucose and insulin concentrations, and postprandial plasma GLP-1, PYY, and ghrelin concentrations. Endpoints also include appetite VAS scores, ad libitum meal consumption, mGITQ scores, vital signs, anthropometric measures, and reports of adverse events, which will be assessed at all clinic visits.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult female or male participants who are 20 to 40 years of age at screening (inclusive)
2. Has a BMI between 18.5 to 29.9 kg·m^(-2) (inclusive) at Visit 1
3. In good general health (no uncontrolled diseases or conditions) as deemed by the investigator and able to consume the study product
4. Individuals with childbearing potential must agree to practice an acceptable form of birth control (i.e., use for at least 3 months prior to the first dose of study product: hormonal contraceptives including oral contraceptives, hormone birth control patch (e.g., Ortho Evra), or hormone implant (e.g., Norplant System); or condoms)
5. Has maintained stable use of medication and supplements defined in the study protocol (Section 7.6), stable dietary and lifestyle habits, and stable body weight, for the last 3 months prior to screening and agree to maintain them throughout the study
6. Agree to avoid strenuous exercise 48 hours prior to each visit
7. Willing to limit daily alcohol consumption to no more than 3 standard drinks per day throughout the study, and agree to entirely avoid alcohol consumption 48 hours prior to each visit (a standard serving is defined here as 4 oz wine, 12 oz beer, 1 oz spirits)
8. Willing to maintain current use of cannabinoids (if applicable) throughout the study
9. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures

Exclusion Criteria:

1. Individuals who are lactating, pregnant or planning to become pregnant during the study
2. Individual with irregular menstrual cycles (defined as outside 24-38 days cycle range, based on self-reports)
3. Individuals who adhere to a diet (e.g., vegan diet) that restricts consumption of dairy products
4. Has a known sensitivity, intolerability, or allergy to any of the study products or their excipients
5. Weight loss or gain > 3 kg in the 3 months prior to Visit 2 (Day 1)
6. Currently or planning to be on a weight loss regimen during the study
7. Received a vaccine for COVID-19 in the two weeks prior to screening or plans to receive a vaccine for COVID-19 during the study period, currently has COVID-19 or tests positive for COVID-19 within 28 days prior to baseline visit, or currently has any post COVID-19 condition(s) as defined by World Health Organization (WHO) (i.e., individuals with a history of probable or confirmed SARS-CoV-2 infection, usually three months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis)
8. Recent [within 2 weeks of Visit 2 (Day 1)] history of an episode of acute GI illness such as nausea/vomiting or diarrhea
9. Have a history of irritable bowel disease (IBS), inflammatory bowel disease (IBD, including ulcerative colitis and Crohn's disease), functional constipation or diarrhea (defined by the Rome IV diagnostic criteria), celiac disease, malabsorption, gastroparesis, diverticulosis, gastric or duodenal ulcers, pancreatitis, or eating disorder; or have a history of intestinal surgery (excluding appendectomy or herniorrhaphy) or bariatric surgery
10. Have an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and/or digestion (e.g., history of bowel obstruction)
11. Participated in upper gastrointestinal endoscopy and/or colonoscopy or preparation within 3 months prior to Visit 2 (Day 1)
12. Diagnosed with hypercholesterolemia or hypertriglyceridemia (i.e., elevated fasting low-density lipoprotein (LDL) (≥ 135 mg/dL; ≥ 3.5 mmol/L) or elevated triglycerides (≥ 150 mg/dL; ≥1.7 mmol/L)
13. Has a history of heart disease/cardiovascular disease, uncontrolled hypertension (≥ 140 systolic or ≥ 90 diastolic mmHg), kidney disease (dialysis or renal failure), hepatic impairment or disease
14. Is Type I or Type II diabetic or pre-diabetic [i.e., elevated fasting blood glucose levels (≥ 100 mg/dL; ≥ 5.6 mmol/L) and/or elevated hemoglobin A1c (≥ 6.0%)]
15. Has a history of liver or gallbladder disease or stomach ulcers
16. Has a positive medical history of unstable thyroid disease, previously diagnosed major affective disorder, psychiatric disorder that required hospitalization in the prior year, immune disorders and/or immunocompromised (e.g., HIV/AIDS)
17. Diagnosed with cancer (except localized skin cancer without metastases or in situ cervical cancer) within 5 years prior to the screening visit, or any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential participant at risk because of participation in the study, or influences the results or the potential participant's ability to participate in the study
18. Major surgery in 3 months prior to screening or planned major surgery during the study
19. History of alcohol or substance abuse (including cannabinoids) in the 12 months prior to screening (including having been hospitalized for such in an in-patient or out-patient intervention program)
20. Use of any treatment listed in the study protocol (Section 7.6) outside of the permitted timeframes and/or conditions.
21. Receipt or use of test products in another research study within 30 days prior to Visit 2 or longer if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study
22. Current or previous tobacco use within the last 6 months
23. Self-report of blood donation totaling between 101 mL to 449 mL of blood within 30 days prior to screening or a blood donation of more than 450 mL within 56 days prior to baseline
24. Self-report of donating plasma (e.g., plasmapheresis) within 14 days prior to screening.
25. Any other active or unstable medical conditions or use of medications/supplements/therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Early (0-2 h) postprandial plasma total amino acid concentration incremental area-under-the-curve (P3 - WHEY vs. placebo treatment) | 2 hours
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan, arginine, glutamine, glycine, alanine, serine, glutamic acid, aspartic acid, asparagine, tyrosine, cysteine, proline (combined) (µmol·L^(-1)·120 min)

SECONDARY OUTCOMES:
Early (0-2 h) postprandial plasma essential amino acid concentration incremental area-under-the-curve | 2 hours
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan (combined) (µmol·L^(-1)·120 min)
Early (0-2 h) postprandial plasma branched chain amino acid concentration incremental area-under-the-curve | 2 hours
  Free leucine, isoleucine, valine (combined) (µmol·L^(-1)·120 min)
Early (0-2 h) postprandial plasma leucine concentration incremental area-under-the-curve | 2 hours
  Free leucine (µmol·L^(-1)·120 min)
Total (0-4 h) postprandial plasma total amino acid concentration incremental area-under-the-curve | 4 hours
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan, arginine, glutamine, glycine, alanine, serine, glutamic acid, aspartic acid, asparagine, tyrosine, cysteine, proline (combined) (µmol·L^(-1)·240 min)
Total (0-4 h) postprandial plasma essential amino acid concentration incremental area-under-the-curve | 4 hours
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan (combined) (µmol·L^(-1)·240 min)
Total (0-4 h) postprandial plasma branched chain amino acid concentration incremental area-under-the-curve | 4 hours
  Free leucine, isoleucine, valine (combined) (µmol·L^(-1)·240 min)
Total (0-4 h) postprandial plasma leucine concentration incremental area-under-the-curve | 4 hours
  Free leucine (µmol·L^(-1)·240 min)
Postprandial plasma amino acid concentration, absolute change from baseline to 45 minutes | 45 minutes
  Total amino acids, essential amino acids, branched chain amino acids, leucine (µmol/L)
Postprandial plasma amino acid concentration, baseline-adjusted change from baseline to 45 minutes | 45 minutes
  Total amino acids, essential amino acids, branched chain amino acids, leucine (µmol/L)
Postprandial plasma amino acid concentration, absolute change from baseline to 60 minutes | 60 minutes
  Total amino acids, essential amino acids, branched chain amino acids, leucine (µmol/L)
Postprandial plasma amino acid concentration, baseline-adjusted change from baseline to 60 minutes | 60 minutes
  Total amino acids, essential amino acids, branched chain amino acids, leucine (µmol/L)
Postprandial plasma amino acid maximum concentration | 4 hours
  Total amino acids, essential amino acids, branched chain amino acids, leucine (µmol/L)
Postprandial plasma amino acid time to peak concentration | 4 hours
  Total amino acids, essential amino acids, branched chain amino acids, leucine (minutes)
Postprandial plasma glucose concentration incremental area-under-the-curve | 4 hours
  Plasma glucose (mmol·L^(-1)·240 min)
Postprandial plasma insulin concentration incremental area-under-the-curve | 4 hours
  Plasma insulin (mmol·L^(-1)·240 min)
Postprandial appetite sensation scores | 4.5 hours
  Participants will be asked to complete visual analog scales (VAS) for measurements of appetite sensations at 10 timepoints (t = 0, 30, 60, 90, 120, 150, 180, 210, 240, and 270 min). Five sensations related to appetite are queried by VAS (i.e., "How hungry are you?", "How full are you?", "How satiated are you?", "How strong is your desire to eat?" on a scale from "Not at all" to "Extremely"; and "How much do you think you could (or would want to) eat right now" on a scale from "nothing at all" to "a very large amount"). Outcomes are measured in millimeters (mm) along a 100-mm horizontal line.
Postprandial appetite sensation incremental-area-under-the-curve | 4 hours
  Participants will be asked to complete visual analog scales (VAS) for measurements of appetite sensations at 9 timepoints (t = 0, 30, 60, 90, 120, 150, 180, 210, 240). Five sensations related to appetite are queried by VAS (i.e., "How hungry are you?", "How full are you?", "How satiated are you?", "How strong is your desire to eat?" on a scale from "Not at all" to "Extremely"; and "How much do you think you could (or would want to) eat right now" on a scale from "nothing at all" to "a very large amount"). Responses are measured in mm·240 min.
Total (0-4 h) postprandial plasma glucagon-like peptide 1 incremental-area-under-the-curve | 4 hours
  Plasma glucagon-like peptide 1 (pg ·L^(-1)·240 min)
Total (0-4 h) postprandial plasma peptide YY incremental-area-under-the-curve | 4 hours
  Plasma peptide YY (pg·L^(-1)·240 min)
Total (0-4 h) postprandial plasma ghrelin incremental-area-under-the-curve | 4 hours
  Plasma ghrelin (pg·L^(-1)·240 min)
Ad libitum meal energy intake | 4.5 hours
  The ad libitum test meal will contain 562 kJ per 100 g with 20% energy from protein, 65% energy from carbohydrate, and 15% energy from fat. The participants will be provided with approximately 1 kg of the test meal on a plate with utensils. Participants will be instructed to "eat as much or as little as desired until feeling "comfortably full" within 30 minutes. The meal will be weighed before consumption and remaining contents will be weighed after achieving comfortable fullness to calculate the energy intake. The outcome will be measure in kilojoules (kJ).
5-Item Palatability Questionnaire scores | 4 hours
  Visual analog score (VAS) outcomes are measured in millimeters (mm) along a 100-mm horizontal line. The most positive and most negative ratings are anchored at each end of the line. The VAS statements on palatability include: (1) "Visual appeal". Responses can range from "Good" to "Bad"; (2) "Smell". Responses can range from "Good" to "Bad"; (3) "Taste". Responses can range from "Good" to "Bad"; (4) "Aftertaste". Responses can range from "Much" to "None"; and (5) "Palatability". Responses can range from "Good" to "Bad".
8-Item Modified Gastrointestinal Tolerance Questionnaire scores | 4 hours
  Participants will be asked to complete an 8-item modified Gastrointestinal Tolerance Questionnaire at the conclusion of each aminoacidemia trial (t = 4 hours). Gastrointestinal symptoms including abdominal bloating/distension, burping, gas/flatulence, borborygmus/stomach rumbling, abdominal cramping, reflux (heartburn), nausea, and vomiting, will be ranked on a 4-point scale ranging from "none" to "severe".
Incidence of adverse events | 72 days
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tyler A Churchward-Venne, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University, Currie Gymnasium (Exercise Metabolism and Nutrition Research Laboratory), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Y, Bell ZW, Alhamwi A, Sauvageau B, Malenda D, Gardy S, Krauth-Ibarz T, Hannaian SJ, Correa JA, Gritsas A, Garvey SM, Tinker KM, Abou Sawan S, Morais JA, Churchward-Venne TA. Acute Effects of Oral Microbial Protease Co-ingestion with Whey Protein on Postprandial Plasma Amino Acid Concentrations, Appetite, and Satiety in Healthy Adults: A Randomized, Double-Blind, Placebo-Controlled, Crossover Clinical Trial. J Nutr. 2025 Oct;155(10):3356-3373. doi: 10.1016/j.tjnut.2025.07.006. Epub 2025 Jul 15. PMID 40675336